CLINICAL TRIAL: NCT00000958
Title: A Placebo-Controlled, Phase I, Pilot Clinical Trial to Evaluate the Safety and Immunogenicity of ENV 2-3, a Yeast-Derived Recombinant Envelope Protein of Human Immunodeficiency Virus-1, in Combination With MTP-PE/MF59 in Individuals With HIV Infection (Placebo Patients Receive MF59 Emulsion Only)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Biocine (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: AVEG 103; 11546 (Registry Identifier: DAIDS ES Registry Number); AVEG 103A; AVEG 103B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Recombinant Proteins; Adjuvants, Immunologic; Acquired Immunodeficiency Syndrome; HIV Envelope Protein gp120; AIDS Vaccines; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Biological: MTP-PE/MF59
Biological: Env 2-3

SUMMARY:
To determine the safety and immunogenicity of Env 2-3 in combination with MTP-PE/MF59 adjuvant in adult volunteers with HIV infection.

By vaccinating those who have HIV infection, perhaps the replication (reproduction) of existing viral strains can be suppressed and the asymptomatic period early in the infectious process can be prolonged. One potential way to do this is to boost HIV antigen-specific CD4 responses, which may in turn increase the effectiveness of CD8 killing of HIV infected cells.

DETAILED DESCRIPTION:
By vaccinating those who have HIV infection, perhaps the replication (reproduction) of existing viral strains can be suppressed and the asymptomatic period early in the infectious process can be prolonged. One potential way to do this is to boost HIV antigen-specific CD4 responses, which may in turn increase the effectiveness of CD8 killing of HIV infected cells.

Eight patients are entered in the pilot portion of the study, thirty patients are entered on Part A and fifteen patients are entered on Part B. In the pilot study, patients receive 30 mcg Env 2-3 vaccine plus 0 - 10 mcg MTP-PE/MF59 adjuvant. Patients on Part A receive one of the following: MF59 emulsion only; 100 mcg MTP-PE/MF59 only; 30 mcg Env 2-3 with MF59 emulsion only; or 30 mcg Env 2-3 vaccine with 100 mcg MTP-PE/MF59. Patients on Part B receive either 100 mcg MTP-PE/MF59 only or 30 mcg Env 2-3 vaccine plus 100 mcg MTP-PE/MF59. Treatment is administered on days 0, 28, and 112, and patients are followed for up to 10 months. Per amendment, patients may receive two additional doses of 30 mcg Env 2-3 or placebo in MTP-PE/MF59 at 7 and 10 months (Parts A and B) or 9 and 12 months (Pilot study) after their initial inoculation.

ELIGIBILITY:
Inclusion Criteria

Patients must be:

* Healthy HIV-seropositive adults (generalized lymphadenopathy, seborrheic dermatitis acceptable).
* Negative for HIV plasma culture.
* Available for 6 months follow-up (patients in Pilot study) or 10 months follow-up (patients in Parts A and B).

Prior Medication: Required:

* Part B: Zidovudine (AZT), tolerating a dose of 500 - 600 mg/day for at least 4 months prior to entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Evidence of psychological disorder during the past year that would impair adherence to the protocol.
* Evidence of an AIDS defining opportunistic infection.

Prior Medication:

Excluded:

* Any potential immunomodulating agents (e.g., isoprinosine, imuthiol, lithium) within 90 days of screening.
* Immunosuppressive medications during the past 3 months.
* Part A: Use of zidovudine (AZT) for more than 30 days in the preceding 6 months, or any AZT within the last 30 days.
* Parts A and B: Any non-AZT antiretroviral drug.
* Any other investigational agent within the past 30 days.
* Immunoglobulins within the past 60 days.

Patients may not have the following prior conditions:

* Evidence of psychological disorder during the past year that would impair adherence to the protocol.
* History of an AIDS-defining opportunistic infection.

Use of illicit drugs or significant amounts of alcohol that, in the opinion of the principal investigator, would interfere with compliance with the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8
Dates: Study Completion 1995-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey L, Study Chair
Locations (1):
- Univ. of Rochester AVEG, Rochester, New York, United States

REFERENCES:
- [Background] Keefer MC, Graham BS, McElrath MJ, Matthews TJ, Stablein DM, Corey L, Wright PF, Lawrence D, Fast PE, Weinhold K, Hsieh RH, Chernoff D, Dekker C, Dolin R. Safety and immunogenicity of Env 2-3, a human immunodeficiency virus type 1 candidate vaccine, in combination with a novel adjuvant, MTP-PE/MF59. NIAID AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1996 May 20;12(8):683-93. doi: 10.1089/aid.1996.12.683. PMID 8744579
- [Background] Mohamed OA, Ashley R, Goldstein A, McElrath J, Dalessio J, Corey L. Detection of rectal antibodies to HIV-1 by a sensitive chemiluminescent western blot immunodetection method. J Acquir Immune Defic Syndr (1988). 1994 Apr;7(4):375-80. PMID 8133447